CLINICAL TRIAL: NCT01653652
Title: Mitigation of Seasonal Allergic Rhinitis Symptoms in Adults by Probiotic Intervention
Brief Title: Effect of a Probiotic on Seasonal Allergic Rhinitis Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11.31. NRC
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: grass pollen; allergic rhinitis; TNSS; miniRQLQ
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): maltodextrin powder to be taken daily
  Interventions: Dietary Supplement: Maltodextrin
- Probiotic (Active Comparator): Probiotic blended in maltodextrin powder to be taken daily
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic
Dietary Supplement: Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of the current study is to evaluate the efficacy of administering a probiotic in adult human subjects suffering from allergic rhinitis during seasonal grass pollen exposure.

DETAILED DESCRIPTION:
Adult subjects with documented seasonal allergic rhinitis (SAR) to grass pollen will be assigned to placebo or probiotic groups and take either placebo or probiotic dietary intervention for 8 weeks during the grass pollen allergy season. Total nasal symptom score (TNSS) will be compared over 8 weeks between the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years of age at the time of enrolment.
* Established seasonal allergic rhinitis (clinical history of rhinorrhea, congestion, sneezing, pruritis >2 years)
* Positive Skin Prick Test (SPT)to Grass Pollen (GP).
* Presence of specific IgE to Grass Pollen (GP)
* Have a Body Mass Index in the range 19-32 kg/m2
* Have signed the consent form
* Have been instructed during screening and agreed to not take any probiotic containing products outside the study for the study period

Exclusion Criteria:

* Subjects currently under treatment with antibiotics or undergoing allergen immunotherapy at the time of enrolment
* Pregnancy
* Vasomotor rhinitis, nasal cavity disorders (nasal polyps), ear infections otitis media).
* Other chronic diseases (e.g. gastrointestinal, cardiovascular, infections)
* Subjects diagnosed with asthma
* Subjects currently participating in another interventional clinical trial or having participated in another clinical trial in the last 2 months
* Subjects on chronic use of systemic corticosteroids prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Total nasal symptom score (TNSS) | every day over 8 weeks
  Total nasal symptom score (TNSS) measuring nasal congestion, runny nose, nasal itching and sneezing on a scale of 0-12 will be compared over 8 weeks between the two treatment groups.

SECONDARY OUTCOMES:
Total ocular symptom score (TOSS) | every day over 8 weeks
miniRQLQ | every week for 8 weeks
  Validated rhinoconjunctivitis quality of life questionnaire (mini RQLQ) measured weekly
Individual nasal and ocular symptoms scores | every day over 8 weeks
Well being index | every week over 8 weeks
Medication Score | every week over 8 weeks
Specific IgE | Baseline and end of study

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany